CLINICAL TRIAL: NCT05966818
Title: Assessment of the Renoprotective Effect of Dapagliflozin in Non-Diabetic Patients With Nephrotic Syndrome.
Brief Title: Effect of Dapagliflozin in Non-Diabetic Patients With Nephrotic Syndrome.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amal A. Elkholy, Lecturer of Clinical Pharmacy, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dapagliflozin in NS
Record Dates: First submitted 2023-06-19; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Nephrotic Syndrome
Keywords: Nephrotic Syndrome; SGLT2 inhibitor; dapagliflozin; management; proteinuria
MeSH Terms: conditions — Nephrotic Syndrome; Proteinuria | interventions — dapagliflozin; Standard of Care; Angiotensin-Converting Enzyme Inhibitors

STUDY DESIGN:
Intervention Model Description: The study is a Prospective, Randomized, Interventional, Parallel, Open Label study.
Masking Description: 90 opaque envelopes will be numbered serially and the corresponding letter which denotes the allocation will be put according to the electronic randomization table. Then all envelopes will be closed and put in one box. When the first patient arrives, the envelope will be opened and the patient will be allocated according to the letter inside.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin group and Standard therapy which include either ACEI or ARB (Active Comparator): - The first group (45 patients) will receive Dapagliflozin (Diglifloz) 10 mg orally once daily at any time of day with or without food. Tablets are to be swallowed whole with half a cup of water for 24 weeks and standard therapy which include either angiotensin converting enzyme inhibitor (ACEI) or angiotensin receptor blocker (ARB).
  Interventions: Drug: Dapagliflozin and Standard therapy (ACEI or ARB).; Drug: Standard Therapy (ACEI or ARB).
- Standard therapy which include either ACEI or ARB (Active Comparator): - The second group (45 patients); will receive the standard therapy (ACEI or ARB).
  Interventions: Drug: Dapagliflozin and Standard therapy (ACEI or ARB).; Drug: Standard Therapy (ACEI or ARB).

INTERVENTIONS:
Drug: Dapagliflozin and Standard therapy (ACEI or ARB). — Dapagliflozin (Diglifloz) 10 mg orally once daily for 24 weeks and the standard therapy (ACEI or ARB).
  Other Names: Dapagliflozin (Diglifloz) 10 mg orally once daily and the standard therapy (ACEI or ARB).
Drug: Standard Therapy (ACEI or ARB). — Standard Therapy which include either ACEI or ARB for 24 weeks.
  Other Names: Standard Therapy which include either ACEI or ARB.

SUMMARY:
Dapagliflozin is the first SGLT2 inhibitor to be approved for CKD treatment regardless of diabetes status. Since many etiologies of non-diabetic nephropathy are characterized by intraglomerular hypertension, it was hypothesized that dapagliflozin acutely decreases GFR and proteinuria in patients without diabetes at risk of progressive kidney function loss such as nephrotic patients via a glucose independent hemodynamic mechanism.

The aim of the study is to assess the effect of Dapagliflozin on proteinuria and estimated glomerular filtration rate in non-diabetic patients with nephrotic syndrome in order to slow the decline in kidney function and the progression to ESRD and to prevent the complications of nephrotic syndrome like thrombotic diseases, peritonitis, hyperuricemia, and recurrent infections.

DETAILED DESCRIPTION:
Nephrotic syndrome (NS) is a clinical syndrome defined by massive proteinuria (greater than 40 mg/m2 per hour) responsible for hypoalbuminemia (less than 30 g/L), with resulting hyperlipidemia, edema, and other complications as thrombotic diseases, peritonitis and recurrent infections.

Dapagliflozin is the first SGLT2 inhibitor to be approved for CKD treatment regardless of diabetes status. Since many etiologies of non-diabetic nephropathy are characterized by intra-glomerular hypertension, it was hypothesized that Dapagliflozin decreases GFR and proteinuria in patients without diabetes at risk of progressive kidney function loss via a glucose independent hemodynamic mechanism.

The aim of the study is to assess the effect of Dapagliflozin on proteinuria and estimated glomerular filtration rate in non-diabetic patients with nephrotic syndrome.

The study will include 90 patients with diagnosis of nephrotic syndrome (proteinuria ≥3.5g/24hr, and serum albumin ≤30g/L) and Urine protein/Creatinine Ratio (UPCR) ≥2. Serum creatinine <3mg/dl (265.2umol/L) and eGFR >30 ml/min/1.73 m2. They will assigned randomly into 2 groups. Each group will contain 45 patients.

* The first group will receive Dapagliflozin (Diglifloz) 10 mg orally once daily for 24 weeks and the standard therapy (ACEI or ARB).
* The second group will receive the standard therapy (ACEI or ARB).

A. Baseline assessment:

At baseline , the non-diabetic patients with nephrotic syndrome will undergo:

* A detailed medical history,
* Physical examination,
* Blood pressure,
* Complete blood count (CBC),
* Baseline biochemical laboratory tests including: kidney function tests (Urinary protein/creatinine ratio (UPCR), eGFR, serum albumin, serum creatinine, serum uric acid, Blood urea nitrogen (BUN), lipid profile and serum glucose level

B. Follow up assessment:

Patients will be followed up every four weeks during the study period (6 months) by measuring UPCR, eGFR, serum albumin, serum creatinine, Blood urea nitrogen (BUN), blood pressure, uric acid, glucose level, lipid profile and CBC. In between visits, patients will be contacted via phone for monitoring of any side effects.

C. End of study assessment:

After 6 months, the previous biochemical tests will be performed such as UPCR, eGFR, serum albumin, serum creatinine, Blood urea nitrogen (BUN), blood pressure, uric acid, glucose level, lipid profile and CBC to measure changes from the baseline.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤60 years.
* Patients with diagnosis of nephrotic syndrome (proteinuria ≥3.5g/24hr, and serum albumin ≤30g/L) and Urine protein/Creatinine Ratio (UPCR) ≥2.
* Serum creatinine <3mg/dl (265.2umol/L) and eGFR >30 ml/min/1.73 m2.
* Pathological diagnosis with membranous nephropathy (MN) or focal segmental glomerulosclerosis (FSGS).
* Absence of any contraindication to dapagliflozin (eGFR less than 30).
* On a stable dose of an ACEI or ARB for at least 4 weeks prior to randomization or Initiation of ACEI or ARB.
* Agreed to participate and sign written informed consent.

Exclusion Criteria:

* Diagnosis of type 1 or type 2 diabetes mellitus.
* Autosomal dominant polycystic kidney disease or autosomal recessive polycystic kidney disease or lupus nephritis.
* Active malignancy aside from treated squamous cell or basal cell carcinoma of the skin.
* History of severe hypersensitivity or contraindications to dapagliflozin.
* History of repeated urinary tract infection or fungal infection.
* Patients with Hemodynamic instability or Hypotension.
* History of noncompliance to medical regimens or unwillingness to comply with the study protocol.
* Pregnancy or breastfeeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of the effect of Dapagliflozin on proteinuria. | Change from Baseline UPCR at 6 months
  By measuring UPCR.
Assessment of the effect of Dapagliflozin on proteinuria. | Change from Baseline Serum Albumin at 6 months
  By measuring serum albumin
Assessment of the effect of Dapagliflozin on Glomerular Filtration Rate (GFR). | Change from Baseline Serum Creatinine at 6 months
  By measuring serum creatinine.
Assessment of the effect of Dapagliflozin on Glomerular Filtration Rate (GFR). | Change from Baseline eGFR at 6 months
  By measuring eGFR.

SECONDARY OUTCOMES:
Assessment of the effect of Dapagliflozin on Systolic blood pressure. | Change from Baseline Systolic Blood Pressure at 6 months
  By measuring Systolic blood pressure.
Assessment of the effect of Dapagliflozin on Diastolic blood pressure. | Change from Baseline Diastolic Blood Pressure at 6 months
  By measuring Diastolic blood pressure.
Assessment of the effect of Dapagliflozin on uric acid. | Change from Baseline Uric acid at 6 months
  By measuring uric acid.
Assessment of the effect of Dapagliflozin on lipid profile. | Change from Baseline lipid profile at 6 months
  By measuring lipid profile.

CONTACTS AND LOCATIONS:
Overall Officials: Nagwa A. Sabri, Professor, Study Chair — Department of Clinical Pharmacy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hussein N, Abdelrahman F, Khedr A, Aref H, Halawa MR, ELSharkawy M. Value of Sodium-Glucose Co-Transporter 2 Inhibitor Versus Traditional Medication in Microalbuminuric Diabetic Patients. Curr Diabetes Rev. 2021;17(6):e101120187809. doi: 10.2174/1573399816999201110194413. PMID 33176660
- [Background] Tapia C, Bashir K. Nephrotic Syndrome. 2023 May 29. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK470444/ PMID 29262216
- [Background] Wang CS, Greenbaum LA. Nephrotic Syndrome. Pediatr Clin North Am. 2019 Feb;66(1):73-85. doi: 10.1016/j.pcl.2018.08.006. PMID 30454752
- [Background] Heerspink HJL, Stefansson BV, Correa-Rotter R, Chertow GM, Greene T, Hou FF, Mann JFE, McMurray JJV, Lindberg M, Rossing P, Sjostrom CD, Toto RD, Langkilde AM, Wheeler DC; DAPA-CKD Trial Committees and Investigators. Dapagliflozin in Patients with Chronic Kidney Disease. N Engl J Med. 2020 Oct 8;383(15):1436-1446. doi: 10.1056/NEJMoa2024816. Epub 2020 Sep 24. PMID 32970396